CLINICAL TRIAL: NCT05049317
Title: A Prospective, Multicenter Clinical Study of Preservative Effect on Postoperative Urinary and Sexual Function During Laparoscopic Functional Total Mesorectum Excision for Male Rectal Cancer Patients
Brief Title: Multicenter Study on Postoperative Urinary and Sexual Function During Laparoscopic Functional Total Mesorectum Excision
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: zhengyongbin01
Record Dates: First submitted 2021-09-10; First posted 2021-09-20 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-09

CONDITIONS: Rectal Cancer
Keywords: Rectal Cancer; Nerve plane; Sexual dysfunction; Urinary dysfunction; Total mesorectal excision
MeSH Terms: conditions — Rectal Neoplasms; Sexual Dysfunction, Physiological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FTME group (Experimental): Participants will undergo laparoscopic FTME surgery.
  Interventions: Procedure: Laparoscopic FTME surgery

INTERVENTIONS:
Procedure: Laparoscopic FTME surgery — Nerve plane was defined as the overlying tiny membranous tissue including the nerves, the adipose tissue and the extremely tiny capillaries around the nerve. Following the TME principles, the surgical procedure of FTME was guided by the nerve plane and dissected between the proper fascia of the rectum and nerve plane (the first gap), which could ensure completeness of the nerve plane and the proper fascia of the rectum.

SUMMARY:
Urinary and sexual dysfunctions are among the most common complications in rectal cancer surgery. The aim of this study was to investigate the protective effect of laparoscopic functional total mesorectum excision (FTME) on urinary and sexual function in male patients with mid-low rectal cancer. This is a prospective, single-arm, multicenter, uncontrolled, clinical study in 88 eligible subjects with mid-low rectal cancer. After informed consent, eligible patients will be performed laparoscopic FTME surgery. Patients' demographic, operative detail, postoperative outcomes and follow-up will be recorded prospectively.

DETAILED DESCRIPTION:
Previously, our studies have demonstrated the presence of nerve plane in laparoscopic rectal cancer surgery, which was the overlying tiny membranous tissue including the nerves, the adipose tissue, and the extremely tiny capillaries around the nerve. As a consequence, the concept of nerve plane-oriented functional total mesorectal excision (FTME) was proposed as an optimal surgical procedure about pelvic autonomic nerve preservation in rectal cancer surgery. Following the TME principles, the surgical procedure of FTME was guided by the nerve plane and dissected between the proper fascia of the rectum and nerve plane (the first gap), which could ensure completeness of the nerve plane and the proper fascia of the rectum. This surgical procedure not only ensures radical resection but also protects PAN better, and the investigators also showed the difference between routine TME and FTME in our previous study, which included inferior mesenteric plexus preservation, station 253 nodes dissection, existence of the first gap, Waldeyer's fascia and Denonvillier's fascia (DVF) preservation, neurovascular bundles preservation, and completeness of mesorectum and nerve plane. Currently, it was a lack of higher-level evidence-based evidence to confirm the protective effect of laparoscopic FTME on urinary and sexual function in male patients with mid-low rectal cancer. In the present study, the investigators performed the prospective, single-arm, multicenter, uncontrolled clinical study, eligible patients will be performed laparoscopic FTME surgery. Postoperative sexual function, urinary function, complications, quality of life, recurrence rate, recurrence patterns, disease-free survival, and overall survival will be recorded prospectively. The results of the patients will be assessed to validate postoperative functional outcomes and oncologic outcomes of laparoscopic FTME surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Male, 18-70 years of age, informed consent;
2. Tumors from anal edge 6 ~ 12 cm (measured by rigid proctoscope);
3. Rectal cancer confirmed pathologically by endoscopic biopsy;
4. Preoperative cT1-3aN0M0 stage (ESMO, 2013);
5. Ro resection is expected;
6. Normal urinary function, normal erection function and ejaculation function grading as I level;

Exclusion Criteria:

1. History of abdominal and pelvic major surgery;
2. Emergency surgery is needed due to the complication (bleeding, obstruction, or perforation) caused by rectal cancer;
3. Pelvic or distant metastasis;
4. Neoadjuvant radiotherapy or chemoradiotherapy;
5. No sexual life;

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2021-11-24 (Estimated); Primary Completion 2022-09-24 (Estimated); Study Completion 2028-09-24 (Estimated)

PRIMARY OUTCOMES:
Incidence of sexual dysfunction | 6 months
  The 5-item version of the International Index of Erectile Function (IIEF-5) and ejaculation function are used to assess sexual function. the IIEF-5 total score ranged from 1 to 25, with a lower score indicating more severe erectile dysfunction, male sexual dysfunction was defined as the IIEF-5 score ≤11points. Ejaculation function was classified as: Grade I, normal ejaculation; Grade II: retrograde ejaculation; Grade III: anejaculation, and ejaculation dysfunction was identified as ejaculation function of grade II/III.
Incidence of urinary dysfunction | 3 months
  The International Prostate Symptom Score (IPSS) are used to assess urinary function. the IIEF-5 total score ranged from 0 to 35, with a higher score indicating more severe erectile dysfunction,moderate-to-severe urinary dysfunction was defined as the IPSS score >8 points.

SECONDARY OUTCOMES:
Morbidity | 30 days
  incidence of postoperatvie complications
Mortality | 30 days
  incidence of postoperatvie deaths
3-year overall survival rate | 36 months
  3-year overall survival rate
3-year disease free survival rate | 36 months
  3-year disease free survival rate
5-year overall survival rate | 60 months
  5-year overall survival rate
5-year disease free survival rate | 60 months
  5-year disease free survival rate
Incidence of sexual dysfunction | 12 months
  The 5-item version of the International Index of Erectile Function (IIEF-5) and ejaculation function are used to assess sexual function. the IIEF-5 total score ranged from 1 to 25, with a lower score indicating more severe erectile dysfunction, male sexual dysfunction was defined as the IIEF-5 score ≤11points. Ejaculation function was classified as: Grade I, normal ejaculation; Grade II: retrograde ejaculation; Grade III: anejaculation, and ejaculation dysfunction was identified as ejaculation function of grade II/III.
Incidence of urinary dysfunction | 6 months
  The International Prostate Symptom Score (IPSS) are used to assess urinary function. the IIEF-5 total score ranged from 0 to 35, with a higher score indicating more severe erectile dysfunction,moderate-to-severe urinary dysfunction was defined as the IPSS score >8 points.

CONTACTS AND LOCATIONS:
Overall Officials: Yongbin Zheng, M.D,Ph.D, Principal Investigator — Renmin Hospital of Wuhan University
Locations (1):
- Yongbin Zheng, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li K, He X, Tong S, Zheng Y. Nerve plane: An optimal surgical plane for laparoscopic rectal cancer surgery? Med Hypotheses. 2021 Sep;154:110657. doi: 10.1016/j.mehy.2021.110657. Epub 2021 Aug 5. PMID 34388537
- [Background] Li K, He X, Zheng Y. An Optimal Surgical Plane for Laparoscopic Functional Total Mesorectal Excision in Rectal Cancer. J Gastrointest Surg. 2021 Oct;25(10):2726-2727. doi: 10.1007/s11605-021-05035-9. Epub 2021 Jun 9. PMID 34109532